CLINICAL TRIAL: NCT04132297
Title: Asthma Academy: Use of Simulation and Telehealth to Empower Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Josiah Macy, Jr. Foundation (Unknown)
Responsible Party: Principal Investigator, Cynthia Foronda, Associate Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190884
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Caregiver Burnout
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Asthma Academy Training + Telehealth Visit Group (Experimental): Participants will receive the Asthma Academy Training virtually. One week after the virtual training, participants will be scheduled to complete a Telehealth visit via zoom through their smart phones or computers.
  Interventions: Behavioral: Asthma Academy; Behavioral: Telehealth Visit
- Virtual Asthma Academy Training (Experimental): Participants will receive the virtual Asthma Academy Training via zoom through their smart phones or computers.
  Interventions: Behavioral: Asthma Academy

INTERVENTIONS:
Behavioral: Asthma Academy — The Asthma Academy is a one hour virtual training that includes providing information about asthma, asthma medications, communicating with healthcare providers and navigating healthcare resources.
Behavioral: Telehealth Visit — The telehealth Visit will be conduct by a trained Doctor of Nurse Practice (DNP) student via a scheduled meeting through zoom on the participant's smart phone or computer. The visit will last about one hour wherein participant will be asked about their asthma knowledge and will be given information about asthma.
  Arms: Virtual Asthma Academy Training + Telehealth Visit Group

SUMMARY:
The goal of this project is to implement and evaluate a novel intervention for low-income families to reduce the burden of caregivers of a child with asthma.

ELIGIBILITY:
Inclusion criteria:

1. Must be age 18 or older
2. Able to speak and read English or Spanish
3. Have a smartphone or computer with active service
4. Care for a child with asthma between ages 5-12
5. Agree to participate

Exclusion criteria:

1. Age less than 18
2. Inability to speak and read English or Spanish
3. Does not have a smartphone or computer with active service
4. Child does not have asthma
5. Care for a child less than 5 or greater than 12
6. Decline to participate
7. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver's asthma knowledge | Baseline, Week 3
  The preliminary effect of the intervention in caregiver's asthma knowledge will be assessed via the Asthma Knowledge Questionnaire. The questionnaire is completed by the caregiver and has 17 items with a total score range of 17-85 with a higher score indicating higher asthma knowledge.
Change in Caregiver's sleep | Baseline, Week 3
  The preliminary effect of the intervention in caregiver's sleep will be assessed via the Adult Sickle Cell Quality of Life Measurement (ASCQ-Me) Version 2.0 Sleep Impact - Short Form Questionnaire. The questionnaire is completed by the caregiver and has 5 items with each item having a scoring possibility of 1-5. The total score ranges from 5-25 with a higher score indicating better sleep.
Change in Caregiver's anxiety | Baseline, Week 3
  The preliminary effect of the intervention in caregiver's anxiety will be assessed via the Quality of Life in Neurological Disorders (Neuro-QOL ) Anxiety - Short Form Questionnaire. The questionnaire is completed by the caregiver and has 8 items with each item having a scoring possibility of 1-5. The total score ranges from 8-40 with a higher score indicating increased anxiety symptoms.
Change in Caregiver's depressive symptoms | Baseline, Week 3
  The preliminary effect of the intervention in caregiver's depressive symptoms will be assessed via the Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Depression - Short Form 8a Questionnaire. The questionnaire is completed by the caregiver and has 8 items with each item having a scoring possibility of 1-5. The total score ranges from 8-40 with a higher score indicating increased depressive symptoms.
Performance of DNP students conducting the Teleheath Visits | Week 3
  Performance of the DNP students conducting the telehealth visits will be evaluated by the average score rated by a faculty and a peer for each DNP. Each total score is tallied from 5 performance categories with each category having a scoring possibility of 0-3. The total score ranges from 0-15 with the higher score indicating a better performance.
Correlation of DNP student performance with family caregiver outcome | Week 3
  The correlation of the performance of the DNP student providing the intervention will be evaluated against the caregiver's asthma knowledge, sleep, anxiety and depressive symptom outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Foronda, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foronda C, Prather S, Snowden K, Gonzalez JM, Gattamorta KA, Lee J, Gonzalez JE, Cardenas M. Asthma academy: A student nurse-led telehealth education program for low-income family caregivers of children with asthma. Nurs Open. 2022 Mar;9(2):1486-1496. doi: 10.1002/nop2.1123. Epub 2021 Dec 16. PMID 34913268